CLINICAL TRIAL: NCT06845553
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Groups, Phase 2a Clinical Trial to Explore the Efficacy and Evaluate the Safety of Vutiglabridin in Knee Osteoarthritis Patients Following 26 Weeks of Oral Treatment
Brief Title: A Study to Assess the Efficacy and Safety of Vutiglabridin in Knee Osteoarthritis Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glaceum (Industry)
Collaborators: Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSG4112-P2-02
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis (Knee OA)
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vutiglabridin 600 mg Multiple Dose (Experimental): Multiple oral dosing of Vutiglabridin 600 mg for 26 weeks
  Interventions: Drug: Vutiglabridin
- Vutiglabridin 1000 mg Multiple Dose (Experimental): Multiple oral dosing of Vutiglabridin 1000 mg for 26 weeks
  Interventions: Drug: Vutiglabridin
- Placebo (Placebo Comparator): Multiple oral dosing of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vutiglabridin — Once-daily oral administration
  Other Names: HSG4112,2-(8,8 dimethyl 2,3,4,8,9,10 hexahydropyrano[2,3 f]chromen 3 yl) 5 ethoxyphenol
  Arms: Vutiglabridin 1000 mg Multiple Dose; Vutiglabridin 600 mg Multiple Dose
Drug: Placebo — Once-daily oral administration
  Arms: Placebo

SUMMARY:
1. Study Objective To Explore the Efficacy and Evaluate the Safety of Vutiglabridin in Knee Osteoarthritis Patients
2. Background Glaceum Inc. has evaluated the safety, tolerability, and pharmacokinetic/pharmacodynamic properties of vutiglabridin in healthy subjects through its Phase 1 trials, and is planning to perform this Phase 2a trial to assess the efficacy and safety of vutiglabridin in Knee Osteoarthritis Patients
3. Study Design and Protocol This study is a randomized, double-blind, placebo-controlled, parallel-group trial. Subjects deemed eligible to participate in this study based on the inclusion/exclusion criteria will be assigned a subject number and randomized to one of the 3 treatment groups - 1 group receiving a placebo - in a 1:1:1 ratio. Subjects will be randomized to double-blind treatments and will receive a once-daily oral dose of the investigational product for 26 weeks according to the study protocol. Several parameters (i.e., 100mm VAS, WOMAC pain subscale, X-ray, MRI, BMI) will be evaluated to assess the efficacy of vutiglabridin. Assessments including measurement of vital signs, 12-lead ECG, clinical laboratory test, pregnancy test, physical examination, and adverse event monitoring will be performed to evaluate the safety and tolerability of vutiglabridin. Blood samples will be collected for pharmacokinetic assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agreed to participate in the study after being informed about the nature of the trial and has signed the informed consent form approved by the IRB.
2. Adults aged 40 to 75 years at the time of screening.
3. Meets the American College of Rheumatology (ACR) criteria for osteoarthritis and has symptoms lasting for more than 3 months requiring pharmacological treatment. Must have knee pain and radiographic evidence of osteophytes, with at least one of the following:

   * Age 50 or older
   * Morning stiffness less than 30 minutes
   * Crepitus on knee motion
4. Has a Kellgren-Lawrence grade II or III in the knee joint on X-ray at the time of screening.
5. Experiences a maximum pain of 50 mm or greater on the 100 mm VAS in activity over the past 24 hours at screening and baseline.
6. For females, the following conditions apply:

   * For women of childbearing potential, the serum hCG pregnancy test at screening must be negative, confirming not pregnant.
   * Not currently breastfeeding.
   * Has undergone surgical sterilization (documented bilateral tubal ligation, bilateral tubal occlusion, bilateral oophorectomy, or hysterectomy), or is postmenopausal.

     * Definition of menopause:
   * For women over 50 years: 12 months of natural amenorrhea.
   * For women under 50 years: Serum FSH level over 40 IU/L and 12 months of natural amenorrhea.

Exclusion Criteria:

1. BMI of 35.0 kg/m² or higher at screening.
2. Developed a clinically significant new disease within 4 weeks before screening or during the screening period, as judged by the investigator.
3. Has arthritis in joints other than the knee.
4. Has any other joint disease except knee osteoarthritis (e.g., secondary osteoarthritis due to trauma, congenital defects, calcium deposition diseases, rheumatoid arthritis, gouty arthritis, Paget's disease, systemic inflammatory disorders, chondrocalcinosis, hemachromatosis, inflammatory arthritis, avascular necrosis, etc.).
5. Has a history of knee or other joint surgery.
6. Has received injections in the affected knee before the administration of the study drug:

   * Steroid injections within 3 months (13 weeks) to the knee osteoarthritis area.
   * Short-acting hyaluronic acid injections within 3 months (13 weeks) to the knee osteoarthritis area.
   * Long-acting hyaluronic acid injections within 6 months (26 weeks) to the knee osteoarthritis area.
7. Has received drug therapy for pain control or symptom improvement in the knee joint area within 4 weeks before study drug administration (opioid analgesics, non-opioid analgesics, topical capsaicin, NSAIDs, anticonvulsants, and other treatments like physical therapy, prolotherapy, herbal treatment, glucosamine, chondroitin).
8. Expected to undergo surgery during the clinical trial period that may affect study completion or adherence to the clinical protocol.
9. Has neuropathic pain or has taken neuropathic pain medications (gabapentinoids, SNRIs, tricyclic antidepressants) within 4 weeks before screening.
10. Has a history of myocardial infarction, unstable angina, stroke, transient ischemic attack, or deep vein thrombosis within 3 months (13 weeks) before screening.
11. Has any clinically significant untreated or unstable diseases of the liver, kidney, nervous system, immune system, respiratory system, endocrine system, blood/oncologic diseases, cardiovascular diseases, psychiatric disorders, neoplastic diseases, or any other conditions deemed unsuitable for participation by the investigator.
12. For males, has a history of hypogonadism or known causes of hypogonadism (e.g., prostate cancer treatment), infertility, Klinefelter syndrome, or Kalman syndrome.
13. Has used medications that can alter reproductive hormone levels (e.g., anabolic steroids, androgens, anti-estrogens, glucocorticoids, opiates, etc.) within 6 months (26 weeks) before screening.
14. Has a history of organ transplantation.
15. Has clinically significant liver dysfunction (e.g., AST or ALT more than 2.5 times the upper limit of normal, total bilirubin more than twice the upper limit of normal [except documented Gilbert's syndrome]) or kidney dysfunction (GFR <60 mL/min).
16. Tests positive for HBsAg, HCV Ab, HIV Ag/Ab, or VDRL (RPR) at screening.
17. Has a history of malignant tumors within the past 5 years (except for those with completely treated basal cell carcinoma, in situ carcinoma, thyroid cancer, or squamous cell carcinoma of the skin, based on the investigator's medical judgment).
18. Has used systemic steroids for 7 or more consecutive days within 3 months (13 weeks) before screening.
19. Has taken immunosuppressive drugs including methotrexate or antimetabolites within 3 months (13 weeks) before screening.
20. Taking drugs that are substrates of the breast cancer resistant protein (BCRP) (e.g., rosuvastatin, sulfasalazine) at screening (however, can be eligible if switched to a different drug in the same class).
21. Has a history of alcohol or drug abuse within 2 years before screening or tests positive for substance abuse at screening (except for documented chronic pain treatment with prescribed medications approved by the investigator).
22. Has participated in another clinical trial or bioequivalence study within 6 months (26 weeks) before the first dose and received investigational medicinal products (except for placebo).
23. Has a history of hypersensitivity or allergic reactions to any components of the investigational medicinal product.
24. Has lactose intolerance.
25. Unwilling to use medically acceptable contraception during the clinical trial period and for 90 days after the last dose.

    * Medically acceptable contraception includes:
    * Oral hormonal contraceptives for female partners of male subjects.
    * Intrauterine devices with proven pregnancy failure rate.
    * Surgical sterilization (e.g., vasectomy, tubal ligation, hysterectomy).
26. Unwilling to donate sperm/eggs during the trial or for 90 days after the last dose.
27. Deemed unsuitable for participation in the trial based on clinical laboratory results or other reasons determined by the investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-19 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 100 mm VAS | From baseline to Week 26
  Change from baseline (Day 1) in the maximum pain experienced during daily activity in the past 24 hours, as assessed by the subject using a 100 mm VAS(Visual Analog Scale; 0=no pain, 100=pain as bad as you can imagine) , at Week 26 post-dosing.

SECONDARY OUTCOMES:
Change from baseline in 100 mm VAS | From baseline to Week 4, 8, 13
  Change from baseline (Day 1) in the maximum pain experienced during daily activity in the past 24 hours, as assessed by the subject using a 100 mm VAS(Visual Analog Scale; 0=no pain, 100=pain as bad as you can imagine) , at Week 4,8,13 and 26 post-dosing.
Change from baseline in 100 mm VAS (weight-bearing) | From baseline to Week 4, 8, 13, 26
  Change from baseline (Day 1) in pain experienced during weight-bearing, as assessed by the subject using a 100 mm VAS, at Weeks 4, 8, 13, and 26 post-dosing.
Change from baseline in 100 mm VAS (at rest) | From baseline to Week 4, 8, 13, 26
  Change from baseline (Day 1) in pain experienced at rest, as assessed by the subject using a 100 mm VAS, at Weeks 4, 8, 13, and 26 post-dosing.
Change from baseline in 100 mm VAS (at night) | From baseline to Week 4, 8, 13, 26
  Change from baseline (Day 1) in pain experienced at night, as assessed by the subject using a 100 mm VAS, at Weeks 4, 8, 13, and 26 post-dosing.
Change from baseline in WOMAC pain subscale | From baseline to Week 4, 8, 13, 26
  Change from baseline (Day 1) in the total WOMAC(Western Ontario and McMaster Universities Osteoarthritis Index) score and scores for each subscale (pain, function, and stiffness) as assessed by the subject, at Weeks 4, 8, 13, and 26 post-dosing.
Subjects who reached a score of 30 mm or less on the 100 mm VAS. | From baseline to Week 4, 8, 13, 26
  The proportion of subjects who reached a pain score of 30 mm or less on the 100 mm VAS at Weeks 4, 8, 13, and 26 post-dosing, as assessed by the subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No